CLINICAL TRIAL: NCT01773629
Title: Care Managers for Perinatal Depression (CMPD)
Acronym: CMPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Collaborators: University of Pennsylvania (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010-38-LGH
Record Dates: First submitted 2013-01-16; First posted 2013-01-23 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Depression; Pregnancy
Keywords: Depression; Pregnancy; Postpartum; Perinatal
MeSH Terms: conditions — Depression | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will receive standard care plus the addition of a care manager. Care managers will function to provide culturally competent and linguistically appropriate support for the care of women identified as being at high risk for depression in pregnancy. Working with both the care providers and these study participants care managers will serve as connectors, coaches, collaborators, and negotiators working to overcome barriers to depression care delivery.
  Interventions: Other: Intervention
- Control (Other): Standard of care: within the current care processes, a woman initiating prenatal care completes a depression risk assessment using a two-step approach. Women with high risk of depression are then scheduled for a separate visit with a member of the care team (a physician, psychologist, or other mental health provider) referred to as a "perinatal depression champion" for a timely formal diagnostic interview.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — Participants in the intervention arm will receive standard care plus the addition of a care manager. Care managers will function to provide culturally competent and linguistically appropriate support for the care of women identified as being at high risk for depression in pregnancy. Working with both the care providers and these study participants care managers will serve as connectors, coaches, collaborators, and negotiators working to overcome barriers to depression care delivery.
  Arms: Intervention
Other: Control — Standard of care: within the current care processes, a woman initiating prenatal care completes a depression risk assessment using a two-step approach. Women with high risk of depression are then scheduled for a separate visit with a member of the care team (a physician, psychologist, or other mental health provider) referred to as a "perinatal depression champion" for a timely formal diagnostic interview.
  Arms: Control

SUMMARY:
The investigators will evaluate effects of introducing the care manager on:

1. Patient receipt of timely diagnosis and initiation of treatment for major depression (diagnosis within 2 weeks of screening and treatment within 1 month of diagnosis); and
2. Patient continuity of care for depression across the transition of care from pregnancy to postpartum (within 4 months postpartum).

DETAILED DESCRIPTION:
The first two specific research aims of this proposed randomized study will evaluate the benefits of introducing site specific care managers into established multi-component enhancements of perinatal depression care. The four study sites are members of the IMPLICIT perinatal quality improvement network and provide prenatal care to a diverse population of low income minority women using a common set of care processes within diverse practice models including Obstetric, Family Medicine, and Nurse Practitioner/Midwifery settings. The established processes of care include evidence based screening, diagnosis, treatment protocols and quality improvement care teams.

The investigators will evaluate effects of introducing the care manager on:

1. Patient receipt of timely diagnosis and initiation of treatment for major depression (diagnosis within 2 weeks of screening and treatment within 1 month of diagnosis); and
2. Patient continuity of care for depression across the transition of care from pregnancy to postpartum (within 4 months postpartum).

For the third and fourth specific research aims we will conduct supplementary econometric and qualitative analyses to aid in understanding the provider and system context in which this intervention is implemented across the four study sites. Results of this evaluation will be used to understand for whom and in which systems of care this model is most successful as well as the costs of delivering this intervention.

Specifically the investigators will:

1. Employ econometric techniques to quantify the costs of implementing and maintaining the IMPLICIT collaborative care maternal depression intervention; and
2. Develop institutional ethnographies of the four study sites and identify factors associated with relative success in implementing perinatal depression care managers and improving timely diagnosis, initiation, and continuity of depression care.

Achieving these aims will provide the foundation for dissemination of this innovative approach to perinatal depression care delivery throughout the entire growing IMPLICIT network which now extends across the northeast and mid-Atlantic regions of the US; sites which provide perinatal care for low income minority women in urban, rural, and suburban communities. These sites include prenatal practices in the Robert Wood Johnson Foundation Aligning Forces for Quality initiative, the Healthy York County Coalition which is partnering with us to disseminate this work in their region.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Current pregnancy or experienced pregnancy in the past 6 weeks
* Score >= 12 on PHQ9

Exclusion Criteria:

* < age 13
* Mental illness
* Primary language other than English or Spanish

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of major depression within 2 weeks of screening | 2 weeks after screening
  Patient receipt of timely diagnosis for major depression during perinatal period.
Treatment of major depression within 1 month of diagnosis | 1 month
  Patient receipt of timely initiation of treatment for major depression during the perinatal period.
Transition of care from pregnancy to postpartum | 4 months
  Patient continuity of care for depression across the transition of care from pregnancy to postpartum within 4 months postpartum.

SECONDARY OUTCOMES:
Quantify the costs of implementing a care manager | 3 years
  Employ econometric techniques to quantify the costs of implementing and maintaining the care manager for managing perinatal depression.
Qualitative assessment of success in implementation of perinatal depression care management process. | 3 years
  Develop institutional ethnographies of the study sites and identify factors associated with relative success in implementing perinatal depression care managers and improving timely diagnosis, initiation, and continuity of depression care. Qualitative measures include efficacy of core implementation group, commitment of implementation group, commitment of user group and readiness to change.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ratcliffe, MD, MSPH, Principal Investigator — Lancaster General Hospital; Ian M Bennett, MD, PhD, Principal Investigator — University of Pennsylvania; Donna Cohen, MD, MS, Principal Investigator — Lancaster General Hospital; Michael A Horst, PhD, MPHS, MS, Principal Investigator — Lancaster General Hospital
Locations (4):
- United States (4):
  - Downtown Family Medicine, Lancaster, Pennsylvania
  - Southeast Lancaster Health Services, Lancaster, Pennsylvania
  - Broad Street Health Center, Philadelphia, Pennsylvania
  - Haddington Health Center, Philadelphia, Pennsylvania